CLINICAL TRIAL: NCT03714412
Title: Feasibility Study of High Surgical Risk Patients With Severe Mitral Regurgitation Treated With the Cardiovalve Transfemoral Mitral Valve System
Brief Title: Feasibility Study of Patients With Severe MR Treated With the Cardiovalve TMVR System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Amended and merged with AHEAD-EU study
Sponsor: Cardiovalve Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL008
Record Dates: First submitted 2018-10-07; First posted 2018-10-22 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implantation (Experimental): Eligible patients will undergo implantation with the Cardiovalve system
  Interventions: Device: Implantation

INTERVENTIONS:
Device: Implantation — Implantation of the Cardiovalve transfemoral mitral valve replacement system
  Other Names: Cardiovalve

SUMMARY:
The study will test the safety and performance of the Cardiovalve transfemoral mitral valve replacement system in treating patients with severe mitral regurgitation who are at high risk for open chest surgery. The system is comprised of comprised of: 1) an Implant; 2) a Delivery System (DS); and 3) Accessories that are required for the implantation procedure. the procedure is performed under general anesthesia.

DETAILED DESCRIPTION:
The study will test the safety and performance of the Cardiovalve transfemoral mitral valve replacement system in treating patients with severe mitral regurgitation who are at high risk for open chest surgery. The system is comprised of comprised of: 1) an Implant; 2) a Delivery System (DS); and 3) Accessories that are required for the implantation procedure. The implant procedure is performed under general anesthesia, and the participants will be followed-up at discharge, 1- 3-, 6-, 12- and 24-months post-procedure, in order to check the system functionality and effect on their cardiology status.

ELIGIBILITY:
General Inclusion Criteria:

2. NYHA functional II, III or ambulatory IV 3. Severe mitral regurgitation (MR grade 3-4+) with pronounced secondary MR etiology 4. Subject is on optimal guideline-directed medical therapy for heart failure for at least 30 days or CRT if indicated.

5. Elevated risk for conventional open mitral valve repair or replacement surgery in the consideration of the site Heart Team (including a cardiac surgeon, a cardiologist and imaging specialist as a minimum) based on STS/Euro Score II (per MVARC Part 1), frailty and co-morbidities.

6. Able to undergo Transesophageal Echocardiography (TEE). 7. Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed.

8. The subject commits to return for the scheduled post-operative follow-up visits at the hospital.

Anatomical Inclusion Criteria 9. Suitable for femoral access procedure and trans septal catheterization 10. Native mitral valve geometry and size and LV outflow tract characteristics compatible with the Cardiovalve (as assessed by the independent Screening Committee)

Exclusion Criteria:

Cardiovascular Exclusion Criteria

1. Prior stroke or TIA within 3 months or Modified Rankin Scale ≥4 disability
2. Acute myocardial infarction within the previous 30 days
3. Any prior heart valve surgery or transcatheter mitral intervention
4. Any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 30 days
5. Rheumatic heart disease or endocarditis within the previous 3 months
6. Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology
7. Existence of inferior vena cava filter or atrial septal device (contraindicating femoral access and transseptal catheterization)
8. Untreated clinically signiﬁcant coronary artery disease requiring revascularization
9. Tricuspid valve disease requiring surgery or severe tricuspid regurgitation
10. Aortic or pulmonic valve disease requiring surgery
11. CRT/ICD implant within 30 days Anatomical Exclusion Criteria (assessed by pre-procedural imaging)
12. Left Ventricular Ejection Fraction (LVEF) <30%
13. LV end diastolic diameter > 70mm
14. Significant abnormalities of the mitral valve and sub-valvular apparatus.
15. Severe mitral annular or leaflets calcification
16. Left atrial or LV thrombus or vegetation
17. Severe right ventricular dysfunction
18. Severe tricuspid or aortic valve disease

    General Exclusion Criteria
19. Subject who is currently participating in an investigational study, other than this study
20. Hemodynamic instability defined as systolic pressure < 90mmHg or the need for inotropic support or intra-aortic balloon pump or other hemodynamic support device, or any mechanical heart assistance
21. Subject has contrast agent hypersensitivity that cannot be adequately pre-medicated, has an allergy to Nitinol alloys (nickel and titanium), or has intolerance to antiplatelet, anticoagulant, or thrombolytic medications
22. Bleeding diathesis or hypercoagulable state
23. Active peptic ulcer or active gastrointestinal bleeding
24. Pulmonary artery systolic pressure >70 mmHg
25. Patients with renal insufficiency (creatinine > 2.5 mg/dL)
26. Need for emergent or urgent surgery for any reason or any planned cardiac Surgery within the next 12 months
27. Subject with hepatic insufficiency
28. Subject has a co-morbid illness that may result in a life expectancy of less than one year
29. Active infection that requires antibiotic therapy
30. Subject is pregnant, breastfeeding or intend to become pregnant within one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09 (Estimated); Primary Completion 2019-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Freedom from major device- or procedure- related serious adverse events | 30 days
  Evaluate the safety of the Cardiovalve with its associated procedure

SECONDARY OUTCOMES:
Technical success of delivery and deployment of the device | Intraoperative
  Technical success of delivery and deployment of the device in the correct position and retrieval of delivery catheter, without significant mitral stenosis
Freedom from emergency surgery or reintervention | 30 days
  Freedom from emergency surgery or reintervention related to the device or access procedure
Freedom from rehospitalizations or reinterventions due to the underlying condition | 30 days, 3 Months, 6 Months, 12 Months, and 24 Months
  Freedom from rehospitalizations or reinterventions for the underlying condition (e.g., mitral regurgitation, worsening of heart failure)
Reduction in MR grade | 30 days, 3-, 6-, 12 and 24-months
  Reduction in MR grade to either optimal (0+ to trace) or acceptable (reduced by at least 1 grade from baseline with no more than 2+ MR) Number of patients with reduction in MR grade from baseline
NYHA class | 30 days, 3-, 6-, 12 and 24-months
  Improvement from baseline in NYHA functional class; Number of patients with improvement in NYHA class
6 minute walk test | 30 days, 3-, 6-, 12 and 24-months
  Increase in distance from baseline
Improvement in quality of life from baseline | 30 days, 3-, 6-, 12 and 24-months
  Improvement from baseline in quality-of-life (Kansas City Cardiomyopathy Questionnaire improvement by ≥ 10)

CONTACTS AND LOCATIONS:
Locations (2):
- Hygeia Hospital, Athens, Greece
- Silesian Center for Heart Diseases, Zabrze, Poland

IPD SHARING:
Plan to Share IPD: No